CLINICAL TRIAL: NCT01196546
Title: Multi-center, Open-label, 24-week Study to Demonstrate the Efficacy and Safety of Combination Therapy of Vildagliptin/Metformin 50/500 or 50/1000 mg Twice Daily in Patients With T2DM Inadequately Controlled With Metformin
Brief Title: Efficacy and Safety of Combination Therapy of Vildagliptin/Metformin in Patients in Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLMF237ATH01
Record Dates: First submitted 2010-08-28; First posted 2010-09-08 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; vildagliptin; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Metformin

ARMS (1):
- Vildagliptin/metformin (Experimental)
  Interventions: Drug: vildagliptin/metformin

INTERVENTIONS:
Drug: vildagliptin/metformin

SUMMARY:
This study will assess the efficacy and safety of combination therapy of vildagliptin/metformin in patients with T2DM inadequately controlled with metformin 1,000 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes mellitus patients who are treated with metformin monotherapy 1,000 mg daily for at least 3 months
* The patient is required to have HbA1c 6.5-11.0%
* BMI in the range of 22-48 kg/m2

Exclusion Criteria:

* Severe or uncontrolled Type 2 diabetes mellitus (HbA1c> 11.0%)
* Acute metabolic diabetes complications such as ketoacidosis or hyperosmolar state (coma) within the past 6 months
* Congestive heart failure requiring pharmacologic treatment
* Any of following within past 6 months: (1) myocardial infarction; (2) unstable angina (3) coronary artery bypass surgery or percutaneous coronary intervention
* Liver disease such as cirrhosis or chronic active hepatitis

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
HbA1c reduction | 24 weeks after treatment

SECONDARY OUTCOMES:
Proportion of patients who achieve target of HbA1c<6.5% at the end of study | 24 weeks after treatment
To evaluate the effect of combination therapy of vildagliptin (50 mg) plus metformin (500 or 1000 mg) twice daily on FPG and BMI, safety and tolerability profiles | 24 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (8):
- Thailand (8):
  - BMA Medical College and Vajira Hospital, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phamongkutklao Hospital, Bangkok
  - Police General Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Khon Kaen Hospital, Khon Kaen
  - Fort Suranaree Hospital, Nakhon Ratchasima
  - Maharat Nakhon Ratchasima Hospital, Nakhon Ratchasima